CLINICAL TRIAL: NCT04824547
Title: Bel Ağrılı Bireylerde Egzersizlerin Uzun Dönem Devamlılığının Değerlendirilmesi
Brief Title: Evaluation of Long-Term Continuity of Exercises in Low Back Pain Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muzeyyen Oz, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 19/602
Record Dates: First submitted 2021-03-21; First posted 2021-04-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Chronic Low-back Pain
Keywords: exercise; pain; yoga; function
MeSH Terms: conditions — Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization exercise group (Active Comparator): Spinal stabilization exercise will be applied all patients accompanied by physiotherapist.
  Sessions will be included selected exercises according to motor learning phases.
  Interventions: Other: exercise
- yoga group (Active Comparator): Yoga program will be applied all patients in this group accompanied by physiotherapist. Sessions will be included selected breathing exercises, warm up, asana and relaxation.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — All exercises programs will applied two sessions per week, totally eight week..

SUMMARY:
Identification of the long term effects of exercises in individuals with low back pain.

DETAILED DESCRIPTION:
Individuals with low back pain who will participate in the study will be divided into two groups. In the stabilization exercise group will be instructed to perform spinal stabilization exercises and in the yoga group will be instructed to perform yoga program consisting of breathing, relaxation and flexibility exercises. The intensity of the pain will be evaluated through visual analog scale, functional status and quality of life will be evaluated through Oswestry Disability Index(ODI), Nottingham Health Profile (NHP), respectively. The exercise adherence will evaluated Exercise Adherence Rating Scale (EARS). The time-distance characteristics of the gait will be evaluated by the OPTOGAIT photoelectric cell (OPTOGait, Microgate, Italy, 2010) and the treadmill system. Assessments will be repeated before, after the treatment, 6 and 12 month follow-up. Also,the number of back pain attacks of the individuals will be questioned and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Must be low back pain at least 3 months
* Must be visual analog scale rating 3 or more

Exclusion Criteria:

* History of any lumbar spine surgery
* Severe/progressive scoliosis
* Spinal stenosis
* Spondylolisthesis
* Cancer
* Diabetes
* Metabolic syndrome
* History of exercise programs or yoga at least 12 weeks before the onset of study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in pain severity | change from baseline in pain intensity at 8 weeks, 6 and 12 month follow-up.
  Patients' average pain intensities will be assessed by Visual Analog Scale (VAS). Participants asked to mark the intensity of pain on a 10 cm long line, explaining that the leftmost of the line does not have pain, that the pain increases while moving to the right, and that the pain is unbearable on the far right.
Changes of functional status | change from baseline in functional status at 8 weeks, 6 and 12 month follow-up.
  Patient's pain related functional status will be measured by Oswestry Disability Index. The scale is considered the 'gold standard' of low back functional outcome tools. This scale contain questions related to functional activities of pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and traveling. The total score is between 0 and 100. The higher the score, the higher the level of disability.

SECONDARY OUTCOMES:
Changes in quality of life | Change from baseline in life quality levels at 8 weeks, 6 and 12 month follow-up.
  Health-related quality of life will be assessed by Nottingham Health Profile (NHP). The NHP contain 38 questions in 6 subareas: pain, physical abilities, energy level, sleep, social isolation and emotional reaction. The scores range from 0 to 100, with each question assigned a weighted value; the sum of all weighted values in a given sub-area adds up to 100. Lower scores denoting a better quality of life.
Changes in Exercise Compliance | Change from baseline in exercise compliance at 8 weeks, 6 and 12 month follow-up.
  Exercise Adherence Rating Scale (EARS) will be used to evaluate the exercise compliance of individuals. The result score of the questionnaire is between 0 and 64. A higher score indicates greater compliance with exercise.
Changes in the gait | Change from baseline in gait at 8 weeks, 6 and 12 month follow-up.
  The gait of individuals will be evaluated by the valid and reliable OPTOGait photoelectric cell and the treadmill system. The gait of individuals on flat ground at their own pace will be recorded for 1 minute. The effects of the exercises on gait will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Muzeyyen OZ, MSc, Principal Investigator — Hacettepe University; Ozlem ULGER, Proffessor, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akhtar MW, Karimi H, Gilani SA. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial. Pak J Med Sci. 2017 Jul-Aug;33(4):1002-1006. doi: 10.12669/pjms.334.12664. PMID 29067082
- [Background] Saper RB, Lemaster C, Delitto A, Sherman KJ, Herman PM, Sadikova E, Stevans J, Keosaian JE, Cerrada CJ, Femia AL, Roseen EJ, Gardiner P, Gergen Barnett K, Faulkner C, Weinberg J. Yoga, Physical Therapy, or Education for Chronic Low Back Pain: A Randomized Noninferiority Trial. Ann Intern Med. 2017 Jul 18;167(2):85-94. doi: 10.7326/M16-2579. Epub 2017 Jun 20. PMID 28631003
- [Background] Zhu F, Zhang M, Wang D, Hong Q, Zeng C, Chen W. Yoga compared to non-exercise or physical therapy exercise on pain, disability, and quality of life for patients with chronic low back pain: A systematic review and meta-analysis of randomized controlled trials. PLoS One. 2020 Sep 1;15(9):e0238544. doi: 10.1371/journal.pone.0238544. eCollection 2020. PMID 32870936
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220